CLINICAL TRIAL: NCT03004937
Title: Early Auditory Referral in Primary Care (EAR-PC)
Brief Title: Early Auditory Referral in Primary Care
Acronym: EAR-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Philip Zazove, Chair of the Department of Family Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HUM00082363
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-Arm, Non-Randomized, Stepped Wedge (Experimental): All patients who meet the inclusion criteria will receive the same intervention.
  Interventions: Other: Family Medicine Hearing Loss Best Practice Alert

INTERVENTIONS:
Other: Family Medicine Hearing Loss Best Practice Alert — A Best Practice Alert, or BPA, was created in the electronic medical record system, which fires when patients meet the inclusion criteria. It reminds providers to ask their patients if they think have a hearing loss and allows them to respond as needed (refer to audiology, add hearing loss to the problem summary list, or dismiss for one year).

SUMMARY:
Busy Primary Care providers (PCPs) have complex practices with many competing demands, making it difficult to improve their HL identification rates. Little research has been conducted to identify effective approaches to address the poor PCP knowledge and provide tools for them to better identify/refer patients with HL for appropriate intervention. Current data suggests there is a critical need to redesign how PCPs deliver hearing health care (HHC) by developing focused educational programs and simple clinical management tools to help them integrate HHC into their practices. To address this need, this study will educate providers on hearing loss (HL) screening/treatment as well as create a Best Practice Alert (BPA), or clinical prompt, that is configured for maximal effectiveness in reminding PCPs to ask their patients if they think they have a HL. This combination of education for providers and clinical reminder could help increase HL screening rates but how much is not clear. This 5 year R21/R33 study funded by National Institute of Deafness and Communicative Disorders seeks to provide detailed understanding of both how educating providers on HL and the use of an effective BPA affects HL screening rates and identification for people with mild to moderate hearing loss.

DETAILED DESCRIPTION:
The Best Practice Alert (BPA) was developed via an iterative process during a two year pilot phase at one site at each health system. First, a "standard" BPA was developed to be launched at each site during the pilot phase. Similarly, a pilot 10-minute education system was developed to be presented just before the above BPA was launched. Pre and post surveys of clinicians were conducted to evaluate the effectiveness of the education program. After clinicians had experience with the BPA, Cognitive Task Analyses (CTAs) with clinicians were conducted to identify ways to make the BPA more effective, and then the BPA was iteratively improved. Similarly, the CTAs helped the investigators understand why clinicians do or do not use BPAs in general. Using this process, a highly rated, easy to use BPA was created and will be utilized in the actual study. The investigators also revamped the education program to a 10 minute video that focused on clinicians mental models of HL, to be used in the actual study. The bigger study, i.e., the R33 phase, will launch at several Family Medicine practices within each of the two different health systems. One of these systems is a traditional academic institution with only academic faculty (physicians and audiologists), midlevels and residents, and the other is a newer academic system, based within a private health system, that includes non-academic physicians and private audiologists. Patients who trigger the BPA will be 55 years or older, do not have an open referral in their chart to audiology, and do not have a known hearing loss already on their problem summary list (PSL). These patients are asked to complete a Hearing Handicap Inventory (HHI) at check-in, a common hearing loss screening tool (score of 10+ indicates probable hearing loss); the results of this will not be shared with clinicians. If the physician chooses to address the prompt during the patient encounter, the BPA design allows them to, 1) Indicate that the patient declines hearing screening (BPA is dismissed for 1 year), 2) Indicate that the patient already has a known hearing loss (HL) and add HL to the PSL (The BPA will be permanently dismissed), 3) Indicate that the patient does not have any HL at this time (The BPA is dismissed for one year), or 4) refer the patient to audiology for hearing screening. The data generated by the BPA is extracted from the electronic health record (EHR) and analyzed to determine if HL screening rates improve when compared to baseline data, whether or not providers are interacting with the BPA, and whether HL is being added to the PSL. The HHI results are used as the "gold standard," i.e., when compared to the data generated by the BPA, indicate whether or not patients with probable HL are getting appropriate care. When an enrolled patient shows up in Audiology the audiologist is asked to complete a three question survey to verify that 1) the referral was appropriate, 2) what is the severity of hearing loss if any, and 3) were hearing aids recommended. This step is to study whether the BPA is generating appropriate referrals. 20% of patients that score 10 or above on their HHI and/or were referred to audiology are contacted by phone and researchers ask them questions about any conversation they may recall related to HL at their appointment as well as their experience in audiology. Iterative improvements will be made to the BPA based on Cognitive Task Analysis (CTA) interviews with randomly selected providers (mostly family physicians). Finally, the implementation of the BPA into clinical practice is observed using the principles of Normalization Process Theory (NPT) to study whether there are other potential issues that may impact whether patients at risk for HL are being screened and referred. The revamped educational video will be shown a week prior to the BPA going live at each site, and repeating the pre and post evaluations. The investigators will be studying whether the education video increases identification and referral of patients at high risk for HL.

ELIGIBILITY:
Inclusion Criteria:

-55 years or older, doesn't have a known hearing loss on their problem summary list (found in the electronic health record), doesn't already have an open referral to audiology in their chart, and has an encounter with a provider at a participating Family Medicine clinic.

Exclusion Criteria:

- None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Increase in Screening Referrals for Hearing Testing of Patients at High Risk for Hearing Loss | Analysis will be done 3 months after data collection completion to allow time for patients to follow up with audiology.
  Baseline data on providers and the clinics will be compared to post-intervention data to determine if hearing loss screening referrals improved; Investigators will also do a step-wedged analysis to look at differences between clinics that have gone live with the BPA and those who have not yet gone live.

SECONDARY OUTCOMES:
Increase in identification of patients with hearing loss | Analysis will be done 3 months after data collection completion to allow time for patients to follow up with audiology.
  Baseline data on providers will be compared to post-intervention data to determine if the percentage of patients with hearing loss on the problem lists is approaching accepted population rates for this age group

CONTACTS AND LOCATIONS:
Overall Officials: Philip Zazove, MD, Principal Investigator — University of Michigan
Locations (10):
- United States (10):
  - Dominos Farms Family Medicine, Ann Arbor, Michigan
  - Chelsea Family Medicine, Chelsea, Michigan
  - Dexter Health Center, Dexter, Michigan
  - Livonia Health Center, Livonia, Michigan
  - Beaumont Rochester Hills Family Physicians, Rochester Hills, Michigan
  - Beaumont East Area Family Practice, Roseville, Michigan
  - Beaumont Shorepointe Family Physicians, Saint Clair Shores, Michigan
  - Beaumont Family Practice, Saint Clair Shores, Michigan
  - Clearwater Family Medicine, Washington, Michigan
  - Ypsilanti Health Center, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: Yes
In process of data collection. Data will be analyzed, papers written, and results posted in clinicaltrials.gov.